CLINICAL TRIAL: NCT06748898
Title: Effect of Transcutaneous Electrical Nerve Stimulation Based on Wrist-ankle Acupuncture Theory on EC50 of Remifentanil Inhibiting Cardiovascular Response After Tracheal Intubation Under General Anesthesia
Brief Title: Effect of Transcutaneous Electrical Nerve Stimulation Based on Wrist-ankle Acupuncture Theory on EC50 of Remifentanil Inhibiting Responses to Tracheal Intubation Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, Associate Chief Doctor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: TENS-WAA
Record Dates: First submitted 2024-12-15; First posted 2024-12-27 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2024-12

CONDITIONS: Perioperative Analgesia; General Anaesthesia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- T group (Experimental): Patients received TENS-WAA with current stimulation
  Interventions: Other: TENS-WAA
- C group (Sham Comparator): Patients received TENS-WAA without current stimulation

INTERVENTIONS:
Other: TENS-WAA — Before anesthesia induction, two paired of electrode pads will be placed on the upper area 1 and 2 with the skin of the treatment area exposed, and the upper and lower juxtaposition method will be adopted. The electrodes were placed close to the skin and connected with TENStem eco basic (Wuxi Jiajian Medical Device Co., Ltd.). Upper area 2 is at the middle of the palmar side of the forearm, between the palmaris longus and flexor carpi radialis.Upper area 1 is between the ulnar border on the little finger side and the flexor carpi ulnaris tendon.Stimulation parameters of TENS-WAA are alternating dense-disperse wave with a frequency of 2Hz and a pulse width of 200μs, and a frequency of 100Hz with a pulse width of 150μs, alternating every 3 seconds ，intensity required to reachthe maximum tolerable level without causing pain, continuous stimulation until the end of surgery.
  Arms: T group
Other: non TENS-WAA — Before anesthesia induction, two paired of electrode pads will be placed on the same position without current stimulation.

SUMMARY:
During endotracheal tube insertion under general anesthesia, sympathetic nerve activity increases, which leads to increased heart rate, increased blood pressure, and increased catecholamine levels in the blood. It is important for patients to maintain hemodynamic stability during anesthesia induction and ultimately mitigate the cardiovascular stress response associated with tracheal intubation.

Transcutaneous Electrical Nerve Stimulation based on Wrist-Ankle Acupuncture theory (TENS-WAA) is a non-invasive pain treatment method, It has the advantages of easy wearing, concentrated treatment site, safe treatment and needle-free. To date, due to the lack of large-scale clinical use of TENS-WAA, only a few studies have reported the use of TENS-WAA for postoperative pain rehabilitation, especially for perioperative pain management. The aim of this study is to evaluate the median effective dose (ED50) of TENS-WAA for remifentanil inhibiting responses to tracheal intubation under general anesthesia, and to provide a reliable basis for its clinical promotion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-64 years old;
* ASA grade I-Ⅲ;
* BMI≤30kg/m2.

Exclusion Criteria:

* Patients predicted to have difficult airways or those experiencing unsuccessful intubation processes;
* Individuals with psychiatric disorders, cognitive impairments, or other conditions that preclude cooperation;
* Patients who have received acupuncture treatment within the past three months or are undergoing routine acupuncture therapy;
* Individuals with a history of severe cardiovascular disease, hyperthyroidism, or asthma;
* Patients with contraindications to transcutaneous electrical nerve stimulation (TENS), including those with pacemakers, metallic implants, allergies to surface electrodes, skin sensory disorders, skin lesions, scars, or unhealed adhesions.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-02-06 (Actual); Primary Completion 2025-11-14 (Actual); Study Completion 2025-11-14 (Actual)

PRIMARY OUTCOMES:
the half maximum effective concentration (EC50) of remifentanil | The remifentanil concentration was recorded for 2 minutes after successful tracheal intubation.
  Dixon's up-and-down method was used to determine the remifentanil concentration, starting from 3.0 ng/mL (step size of 0.2 ng/mL). After obtaining 7 infection points from positive to negative endotracheal intubation reactions, patient recruitment was terminated. A positive response to endotracheal intubation was defned as MAP 15% above the basal level or HR 15% above the basal level within 2 min of endotracheal intubation. The EC50 of remifentanil Ce was determined by calculating the average of the midpoint dose of all independent pairs of patients after six crossover points were obtained.

SECONDARY OUTCOMES:
The time required for tracheal intubation | The time consumed by this procedure was recorded from the beginning of intubation until completion of inflation of the endotracheal tube cuff
  defined as the time from the start of intubation to inflation of the bronchial tube cuff
Nausea and vomiting | 24 hour after surgery
  Postoperative nausea and vomiting was assessed by visual analogue scale (VAS) : a 10-cm ruler was used as a scale, with 0 at one end indicating no nausea and vomiting, and 10 at the other end indicating the most severe nausea and vomiting that could not be tolerated (1-4 as mild, 5-6 as moderate, 7-10 as severe).
The dynamic VAS score | 24 hour after surgery
  Independent investigators will assess the postoperative dynamic pain (pain during activities or coughing) by utilizing a visual analogue scale (VAS) ranging from 0 to 10. The two ends of the straight line represent "no pain at all" and "the worst pain imaginable," respectively. Patients are required to mark their corresponding position on the line based on their perception of pain, and the numerical value corresponding to this position serves as the patient's pain score.
QoR-15 questionnaire | 24 hour after surgery
  The 15-item QoR score is used to asses quality of recovery after surgery which ranges 0-150 and higher QoR-15 scores indicate better postoperative recovery
Postoperative airway complications | 24 hour after surgery
  Postoperative airway complications such as hoarseness, sore throat, and difficulty in pronunciation are assessed by researchers during postoperative follow-up visits to check for the presence of related complications and to record the findings
Postoperative static pain (pain at rest) | 24 hour after surgery
  Postoperative static pain (pain at rest) will be quantified by utilizing a visual analogue scale (VAS) ranging from 0 to 10. The two ends of the straight line represent "no pain at all" and "the worst pain imaginable," respectively. Patients are required to mark their corresponding position on the line based on their perception of pain, and the numerical value corresponding to this position serves as the patient's pain score.

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Yangpu, China